CLINICAL TRIAL: NCT01974297
Title: Comparison of the Efficacy and AtorVastatin 20mg mOnotherapy Versus Combination Atorvastatin/Fenofibric Acid 10/135mg in the Mixed hyperlipiDemia Who Were Not at Lipid gOals With Atorvastatin 10mg Monotherapy.
Brief Title: Comparison of the Efficacy and Safety of AtorVastatin mOnotherapy vs. Combination Atorvastatin/Fenofibric Acid
Acronym: AVOCADO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sang Hak Lee (Other)
Responsible Party: Sponsor-Investigator, Sang Hak Lee, Associate Professor in Cardiology(preventive cardiology) in Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, Korea, Yonsei University
Organization: Yonsei University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVOCADO
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Mixed Hyperlipidemia
Keywords: Hyperlipidemia; Atorvastatin; Fenofibric acid; combination; monotherapy
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipidemias | interventions — Atorvastatin; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 20mg, monotherapy (Active Comparator): Atorvastatin 20mg/day PO for 12weeks
  Interventions: Drug: atorvastatin 20mg
- Atorvastatin 10mg, Fenofibric acid 135mg (Experimental): Atorvastatin 10mg, Fenofibric acid 135mg per day PO for 12weeks
  Interventions: Drug: Atorvastatin 10mg, fenofibric acid 135mg

INTERVENTIONS:
Drug: Atorvastatin 10mg, fenofibric acid 135mg — Atorvastatin 10mg, fenofibric acid 135mg/day PO for 12 weeks
  Other Names: Newvast 10mg, Fenocid 135mg
  Arms: Atorvastatin 10mg, Fenofibric acid 135mg
Drug: atorvastatin 20mg — Atorvastatin 20mg/day PO for 12weeks
  Other Names: Newvast Tab. 20mg
  Arms: Atorvastatin 20mg, monotherapy

SUMMARY:
The purpose of this study is to compare combination atorvastatin/fenofibric acid 10/135mg with atorvastatin 20mg monotherapy in the mixed hyperlipidemia who were not at lipid goals with atorvastatin 10mg monotherapy.

DETAILED DESCRIPTION:
Study conduct according to the standard operating procedure

* The sponsor, the investigator, and all other persons involved in the study at the study center or other facilities should conduct the study in accordance with the study protocol, each standard operating procedure, and Korea Good Clinical Pratice.

Data quality control

* In order to ensure the reliability of all study-related data and their appropriate processing, the sponsor will apply quality control to each step of data handling

Monitoring

* In order to confirm that the study is being conducted, recorded and reported according to the study protocol and International Conference on Harmonization Good Clinical Practice(ICH-GCP), the sponsor or CRO will perform monitoring of study procedure. In monitoring, the monitors will cross check the description in the case report form, etc. against study-related records such as source documents to confirm that the description is accurate.

Measures taken to cope with adverse events and reporting procedure

* The investigator should notify the event to the sponsor or Contract Research Organization(CRO) immediately (within around 24 hours) after having noticed the occurence of a serioius adverse event by telephone, fax or E-mail. The investigator should complete and submit an serioius adverse event(SAE) report form containing all information to the Institutional Review Board (IRB).

Data Management

* In this study, data will be collected in electronic Case Report Form(CRF)
* Data validation for missing data will be managed by computer programming and manual check.

ELIGIBILITY:
Inclusion Criteria:

* patients of the age of 20years or older
* patients who have been taking atorvastatin 10mg 1 tab per day for more than 8 weeks before screening
* patients who meet the following criteria

  1. Low density lipoproteins-cholesterol level < 130mg/dL
  2. 150mg/dL < Triglyceride level < 500mg/dL
  3. HDL-cholesterol level < 45mg/dL
* patients who consent for the consent before enrolling the study

Exclusion Criteria:

* Allergic to HMG-CoA reductase inhibitor and fibrates
* uncontrolled Hypertension
* unstable angina, myocardial infarction, transient ischemic attack
* uncontrolled diabetes
* thyroid disease
* myopathy, rhabdomyolysis history
* alcoholic
* chronic diarrhea, gastrointestinal disease
* malignant tumor
* patients who are pregnant
* lactating woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Changes of non-HDL cholesterol | at screening and after 12 weeks
  -change rate : [(12nd week non-High density lipoprotein - baseline non-High density lipoprotein) / baseline non-High density lipoprotein] * 100
levelresponse rate of non-HDL cholesterol level < 130mg/dL | at screening and after 12 weeks
  -Response rate : (subjects who are at less than 130mg/dL of non-High density lipoprotein level / all subjects) * 100

SECONDARY OUTCOMES:
changes of TC,HDL-C,LDL-C,TG,Apo B/A1 | at screening and after 12 weeks
Changes of Glucose, HbA1c, HOMA-IR level | at screening and after 12 weeks
  HOMA-IR index = [fasting serum insulin(uU/mL) * fasting serum glucose(mmol/L)]/22.5
Changes of hs-CRP, adiponectin, resistin level | at screening and after 12 weeks

OTHER OUTCOMES:
changes of BUN/Cr level | at screening and after 12 weeks
Changes of Homocysteine level | at screening and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hak Lee, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Goldberg AC, Bays HE, Ballantyne CM, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Efficacy and safety of ABT-335 (fenofibric acid) in combination with atorvastatin in patients with mixed dyslipidemia. Am J Cardiol. 2009 Feb 15;103(4):515-22. doi: 10.1016/j.amjcard.2008.10.025. Epub 2008 Dec 26. PMID 19195513
- [Result] Jones PH, Goldberg AC, Knapp HR, Kelly MT, Setze CM, Stolzenbach JC, Sleep DJ. Efficacy and safety of fenofibric acid in combination with atorvastatin and ezetimibe in patients with mixed dyslipidemia. Am Heart J. 2010 Oct;160(4):759-66. doi: 10.1016/j.ahj.2010.06.045. PMID 20934572
- [Result] Mohiuddin SM, Pepine CJ, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Efficacy and safety of ABT-335 (fenofibric acid) in combination with simvastatin in patients with mixed dyslipidemia: a phase 3, randomized, controlled study. Am Heart J. 2009 Jan;157(1):195-203. doi: 10.1016/j.ahj.2008.08.027. Epub 2008 Nov 20. PMID 19081418
- [Result] Kishikawa R, M-Horiuti T, Togawa A, Kondoh Y, Janzy PD, Goldblum RM, Kotoh E, Shimoda T, Shoji S, Nishima S, Brooks EG. [Juniper pollen monitoring by Burkard sampler in Galveston, Texas, USA and Japanese cedar pollen counting in Fukuoka, Japan -- introduction of Pan American Aerobiology Association protocol counting technique]. Arerugi. 2004 Jun;53(6):582-8. Japanese. PMID 15247520
- [Result] Jones PH, Davidson MH, Kashyap ML, Kelly MT, Buttler SM, Setze CM, Sleep DJ, Stolzenbach JC. Efficacy and safety of ABT-335 (fenofibric acid) in combination with rosuvastatin in patients with mixed dyslipidemia: a phase 3 study. Atherosclerosis. 2009 May;204(1):208-15. doi: 10.1016/j.atherosclerosis.2008.09.027. Epub 2008 Oct 5. PMID 18996523
- [Result] Filippatos TD. A review of time courses and predictors of lipid changes with fenofibric acid-statin combination. Cardiovasc Drugs Ther. 2012 Jun;26(3):245-55. doi: 10.1007/s10557-012-6394-0. PMID 22592524
- [Result] Chatley P, Badyal DK, Calton R, Khosla PP. Combination therapy of low-dose atorvastatin and fenofibrate in mixed hyperlipidemia. Methods Find Exp Clin Pharmacol. 2007 Apr;29(3):217-21. doi: 10.1358/mf.2007.29.3.1075363. PMID 17520105
- [Result] Davidson MH, Rooney MW, Drucker J, Eugene Griffin H, Oosman S, Beckert M; LCP-AtorFen Investigators. Efficacy and tolerability of atorvastatin/fenofibrate fixed-dose combination tablet compared with atorvastatin and fenofibrate monotherapies in patients with dyslipidemia: a 12-week, multicenter, double-blind, randomized, parallel-group study. Clin Ther. 2009 Dec;31(12):2824-38. doi: 10.1016/j.clinthera.2009.12.007. PMID 20110022
- [Result] Shah HD, Parikh KH, Chag MC, Shah UG, Baxi HA, Chandarana AH, Naik AM, Shah JN, Iyer S, Shah KJ, Goyal RK. Beneficial effects of the addition of fenofibrate to statin therapy in patients with acute coronary syndrome after percutaneous coronary interventions. Exp Clin Cardiol. 2007 Summer;12(2):91-6. PMID 18650989
- [Result] Farnier M, Ducobu J, Bryniarski L. Efficacy and safety of adding fenofibrate 160 mg in high-risk patients with mixed hyperlipidemia not controlled by pravastatin 40 mg monotherapy. Am J Cardiol. 2010 Sep 15;106(6):787-92. doi: 10.1016/j.amjcard.2010.05.005. Epub 2010 Aug 2. PMID 20816118